CLINICAL TRIAL: NCT00142818
Title: A Phase II, Double-blind, Placebo-Controlled, Pilot Trial of the Combination of Modafinil and Naltrexone for the Treatment of Cocaine and Alcohol Dependence
Brief Title: Modafinil and Naltrexone to Reduce Cocaine and Alcohol Dependence
Acronym: Mod-Nal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyle Kampman (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Kyle Kampman, Principal Investigator, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-12756-3; P50DA012756-03 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Alcohol-Related Disorders; Alcoholism; Cocaine-Related Disorders
Keywords: Alcohol Abuse; Cocaine Abuse
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism; Cocaine-Related Disorders | interventions — Naltrexone; Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Naltrexone plus modafinil (Experimental): Nal + Mod
  Interventions: Drug: Naltrexone; Drug: Modafinil
- Naltrexone (Experimental): Nal
  Interventions: Drug: Naltrexone
- Modafinil (Experimental): Mod
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — 150 mg daily for males; 100 mg daily for females
  Other Names: ReVia
  Arms: Naltrexone; Naltrexone plus modafinil
Drug: Modafinil — 400 mg daily
  Other Names: Provigil
  Arms: Modafinil; Naltrexone plus modafinil
Drug: Placebo — 400 mg and/or 100-150 mg placebo pills
  Arms: Placebo

SUMMARY:
Modafinil is a medication that may enhance mood and increase energy in cocaine addicts, which may be useful in preventing cocaine relapse. Naltrexone is a medication that is currently used to treat drug and alcohol addiction. A combination of these two medications may be beneficial in reducing drug and alcohol use in individuals undergoing substance abuse treatment. The purpose of this study is to evaluate the effectiveness of modafinil and naltrexone, alone and in combination, at reducing drug and alcohol use in individuals addicted to cocaine and alcohol.

DETAILED DESCRIPTION:
Cocaine and alcohol addiction are serious health problems with no available medical treatment for preventing relapse. Past research has shown that individuals who are addicted to both cocaine and alcohol typically respond poorly to conventional substance abuse treatment. Little attention has been directed towards how best to treat these individuals. Naltrexone is a medication that is currently used to treat drug and alcohol addiction. It acts by blocking the "high" feeling produced by drugs and alcohol. Modafinil, another medication, enhances mood, increases energy, and improves concentration in people with narcolepsy. Preliminary research has shown that it may produce similar effects to cocaine, thereby potentially countering the symptoms of cocaine withdrawal. Cognitive Behavioral Coping Skills Therapy (CBT), a form of therapy that aims to alter an individual's patterns of behavior and drug use, is also an important component of substance abuse treatment. The purpose of this study is to compare the effectiveness of CBT plus placebo, CBT plus modafinil, CBT plus naltrexone, and CBT plus a combination of modafinil and naltrexone at reducing cocaine and alcohol use in individuals addicted to both substances.

This 14-week study will enroll individuals addicted to both cocaine and alcohol. During a 1-week screening period, potential participants will be required to complete a detoxification program, including stopping all cocaine and alcohol use. Participants will also undergo a physical exam and an electrocardiogram. Blood will be drawn for laboratory tests, and urine tests will be used to screen for the presence of drugs and alcohol. Individuals who complete the screening and meet all study requirements will be permitted to participate in the treatment phase of the study. During the 13-week treatment phase, participants will be randomly assigned to receive modafinil, naltrexone, a combination of modafinil and naltrexone, or placebo. All participants will attend a CBT session once a week. Study visits will take place twice a week. At each visit, a urine test and breathalyzer will be used to screen for the presence of alcohol and drugs. Participants will also complete standardized psychological questionnaires to measure drug and alcohol craving, treatment services received, severity of illness, and withdrawal symptoms. In addition, participants will meet weekly with a nurse practitioner, who will dispense study medications, monitor adverse events, and evaluate the participant's clinical status. A follow-up evaluation will occur 6 months following the end of treatment.

ELIGIBILITY:
4.1 Inclusion Criteria

1. Male and females, 18 years of age or older.
2. Meets DSM-IV criteria for current diagnoses of cocaine and alcohol dependence, determined by the SCID-IV.
3. In the past 30 days, used no less than $200-worth of cocaine and meets the following drinking criteria as measured by the Timeline Followback (TLFB) (Sobell, 1995):

   1. drank within 30 days of intake day,
   2. reports a minimum of 48 standard alcoholic (avg. 12 drinks/wk) in a consecutive 30-day period over the 90-day period prior to starting intake (i.e., a minimum of 40% days drinking), and
   3. has 2 or more days of heavy drinking (defined as 5 or more drinks per day in males and 4 or more drinks per day in females) in this same pre-treatment period.
4. 72 consecutive hours of abstinence from alcohol, determined by self-reports and confirmed by a negative breathalyzer tests, and a Clinical Institute Withdrawal Scale for Alcohol (CIWA-AR) (Sullivan, 1989) score below eight. Subjects will be encouraged to achieve 72 consecutive hours of abstinence, however, subjects who have achieved between 48 and 72 consecutive hours of abstinence will be included with the approval of the principal investigator. We anticipate that these subjects will comprise less than 5% of total enrolled subjects. Subjects will be given 2 additional weeks beyond the screening week to attain the appropriate period of alcohol abstinence prior to randomization.
5. Lives a commutable distance from the TRC and agrees to attend all research visits including follow-up visits.
6. Speaks, understands, and prints in English
7. Ability to give informed consent

Exclusion Criteria

1. Abstinent from cocaine or alcohol for 30 consecutive days prior to signing consent form.
2. Meets DSM IV criteria for dependence on any substance other than cocaine and alcohol (except nicotine), determined by the SCID.
3. Needs treatment with any psychoactive medications including any anti-seizure medications (with the exception of diphenhydramine used sparingly, if necessary, for sleep).
4. Meets current or lifetime DSM-IV criteria for schizophrenia or any psychotic disorder or organic mental disorder. Subject meets current DSM-IV diagnosis of any other clinically significant psychiatric disorder that will interfere with study participation.
5. Has evidence of a history of significant hematological, pulmonary, endocrine, cardiovascular, renal or gastrointestinal disease (including a history of myocardial infarction, mitral valve prolapse, left ventricular hypertrophy, uncontrolled hypertension).
6. Severe physical or medical illnesses such as AIDS, active hepatitis, significant hepatocellular injury as evidenced by elevated total bilirubin levels (>1.3 mg/dl),or elevated levels (over 4.5x normal) of aspartate aminotransferase (AST), and serum glutamic-pyruvic transaminase (SGPT) after the required 3 days of abstinence.
7. Use of an investigational medication in the 30 days prior to randomization.
8. History of hypersensitivity to modafinil or naltrexone
9. Receiving chronic therapy with any drug known to interact adversely with either modafinil or naltrexone including propranolol, phenytoin, warfarin, diazepam
10. Took a monoamine oxidase inhibitor within 30 days of randomization.
11. Is female and tests positive on a pregnancy test, is contemplating pregnancy in the next 6 months, is nursing, or is not using an effective contraceptive method (if relevant). Acceptable methods of contraception include barrier methods (diaphragm or condom with spermicide, female condom), intrauterine progesterone contraceptive system, levonorgrestrel implant, and medroxyprogeterone acetate contraceptive injection, copper IUD, vaginal contraceptive film, cervical cap, contraceptive foam.
12. Current use of an oral contraceptive without other acceptable barrier method of contraception.
13. Received therapy with any opiate substitute (methadone, LAAM, buprenorphine) within 60 days of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2006-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M. Kampman, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ModNal: Nal + Mod
  Naltrexone: 150 mg daily for males; 100 mg daily for females
  Modafinil: 400 mg daily
- Naltrexone and Placebo: Nal
  Naltrexone: 150 mg daily for males; 100 mg daily for females
- Modafinil and Placebo: Mod
  Modafinil: 400 mg daily
- Double Placebo: Placebo
  Placebo: 400 mg and/or 100-150 mg placebo pills
Period: Overall Study
Arm/Group | ModNal | Naltrexone and Placebo | Modafinil and Placebo | Double Placebo
Started | 45 | 40 | 37 | 42
Completed | 28 | 19 | 24 | 20
Not Completed | 17 | 21 | 13 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ModNal | Naltrexone and Placebo | Modafinil and Placebo | Double Placebo | Total
Number analyzed (Participants) | 45 | 40 | 37 | 42 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 40 | 37 | 42 | 164
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 5 | 7 | 14 | 41
  Male | 30 | 35 | 30 | 28 | 123
Region of Enrollment [Number; unit: participants]
  United States | 45 | 40 | 37 | 42 | 164

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use (Measured by Timeline Follow Back and Urine Screen From Week 2-week 14)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: number of cocaine negative urine samples
Arm/Group | ModNal | Naltrexone and Placebo | Modafinil and Placebo | Double Placebo
Number analyzed (Participants) | 45 | 40 | 37 | 42
number of cocaine negative urine samples | 9.3 (8.4) | 7.2 (8.1) | 10.1 (9.4) | 10.5 (9.9)

2. Primary Outcome: Percent Days of Heavy Drinking (Measured by Timeline Follow Back Starting at Week Two Through Week 14
Time Frame: 13 weeks
Measure: Mean (Standard Error); unit: mean percentage of days
Groups:
- Modafinil Plus Naltrexone: Nal + Mod
  Naltrexone: 150 mg daily for males; 100 mg daily for females
  Modafinil: 400 mg daily
Arm/Group | Modafinil Plus Naltrexone | Naltrexone | Modafinil | Placebo
Number analyzed (Participants) | 45 | 40 | 37 | 42
mean percentage of days | 34.7 (4.4) | 35.1 (4.2) | 33.6 (4.2) | 33.8 (4.3)
Statistical Analysis 1: Comparison: Modafinil Plus Naltrexone vs Naltrexone vs Modafinil vs Placebo; Test type: Superiority; p = 0.4, ANOVA

ADVERSE EVENTS:
Arm/Group | ModNal | Naltrexone and Placebo | Modafinil and Placebo | Double Placebo
Serious Adverse Events (participants affected / at risk) | 11/45 | 6/40 | 6/37 | 11/42
Other Adverse Events (participants affected / at risk) | 11/45 | 10/40 | 8/37 | 4/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ModNal (N=45) | Naltrexone and Placebo (N=40) | Modafinil and Placebo (N=37) | Double Placebo (N=42)
Hospitalization (General disorders) | 7 (9) | 3 (3) | 3 (3) | 7 (11)
Exacerbation of cocaine and alcohol (General disorders) | 4 (4) | 2 (2) | 3 (3) | 6 (6)
Depression or Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arrested for Homicide (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ModNal (N=45) | Naltrexone and Placebo (N=40) | Modafinil and Placebo (N=37) | Double Placebo (N=42)
Nausea (Gastrointestinal disorders) | 11 | 10 | 8 | 4
Anxiety (Psychiatric disorders) | 9 | 2 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less